CLINICAL TRIAL: NCT02559700
Title: Optimising Engagement in an Online Brain Training Intervention for Adults Over 50
Brief Title: Online Brain Training Intervention for Over 50s
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Alzheimer's Society (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 188008
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: Healthy Ageing
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain training programme (Experimental): Participants will complete a package of online brain training games focusing on reasoning and problem solving. The intervention will be accessed via a computer. There is no minimum or maximum dosage but participants will be recommended to complete the intervention five times a week. The package takes approximately 10 minutes to complete, depending on individual performance.
  Interventions: Behavioral: Brain training programme

INTERVENTIONS:
Behavioral: Brain training programme — An online package of brain training programmes

SUMMARY:
This study is an open trial investigating the long-term use of an online brain training programme for adults over 50. It will determine whether there is sustained benefit to cognition, and whether this group can be engaged in this form of intervention over a period of 12 months.

DETAILED DESCRIPTION:
This study will evaluate an optimised brain training programme to determine whether it is engaging for older adults and whether it results in improvement or maintenance of cognition over a 12 month period.

The Brain Training intervention

The programme is an updated version of the original 'Brain Test Britain' intervention, which was successfully evaluated in a large previous trial. It consists of a series of games or tests, completed on a computer. Each test is designed to target the participants' reasoning and problem-solving ability, for example by asking them to balance weights on a see-saw or select the 'odd-one-out' from a series of shapes. As the participants progress over the course of the study they will receive increasingly more challenging versions of each test, depending on their performance. The intervention has been updated from the original to improve engagement through improved visuals, more intelligent difficulty setting and a more engaging delivery platform.

The research delivery platform: PROTECT

A novel infrastructure resource has been developed at King's College London within the Maudsley Biomedical Research Unit for Dementia (BRU-D), which provides the opportunity to deliver the intervention to large numbers of older adults. The Platform for Research Online to investigate Cognition and Genetics in Ageing (PROTECT) is an online research tool. PROTECT is currently recruiting a cohort of over 10,000 adults over 50 who are cognitively healthy or have early cognitive impairment. Participants provide demographic and lifestyle information and will complete a battery of validated cognitive assessments annually. The focus of all research conducted through PROTECT is on the prevention of dementia and risk reduction. The optimised brain training intervention will be delivered through this platform. PROTECT has ethical approval from the NHS Research Ethics Service Committee for London Bridge (Ref: 13/LO/1578).

Study Design

Design: 12-month open online clinical trial Participants: 5000 adults over 50 Setting: Intervention delivered at home, online through the PROTECT website

Recruitment

Recruitment will be achieved through the PROTECT site through a national advertisement strategy. This will be accomplished through partnerships with the media and third sector. All participants registered on PROTECT will be invited to take part and provided with the information sheet. Participants will consent through the secure online procedure on the PROTECT site.

ELIGIBILITY:
Inclusion Criteria:

* Over 50,
* Have access to a computer and the internet
* Registered as a participant on the PROTECT website

Exclusion Criteria:

* Established diagnosis of dementia

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4387 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in reasoning ability as measured by the Baddeley Grammatical Reasoning | 12 months

SECONDARY OUTCOMES:
Change in visual memory and learning as measured by the Paired Associate Learning Test | 12 months
Change in reaction time as measured by the Simple and Choice Reaction Test | 12 months
Change in spatial working memory as measured by the Spatial Working Memory Test | 12 months
Change in ability to complete day-to-day activities as measured by the Instrumental Activities of Daily Living scale (part of the Home Care Minimum Dataset) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Corbett, PhD, Principal Investigator — King's College London